CLINICAL TRIAL: NCT04179721
Title: Reducing Behavioral and Psychological Symptoms of Dementia (BPSD) for Acutely-Ill Persons With Alzheimers Disease and Related Dementias Via Patient Engagement Specialists
Brief Title: Reducing Behavioral and Psychological Symptoms of Dementia: Hospital Caregivers (Aim 2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Penn State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 19-0800-FIMR-2; 1R21NR018500-01 (NIH)
Record Dates: First submitted 2019-11-20; First posted 2019-11-27 (Actual); Results first posted 2022-10-27 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Alzheimer's Disease and Related Dementias
Keywords: Behavioral and Psychological Symptoms of Dementia; Alzheimer's Disease and Related Dementias; Hospitalization
MeSH Terms: conditions — Alzheimer Disease; Behavior

STUDY DESIGN:
Intervention Model Description: Nonrandom preliminary efficacy trial comparing 2 groups, intervention and control
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The PES-4-BPSD Model (Experimental): The intervention arm consists of PES and NAs who work on the intervention unit which consists of: I. Cohorting of patients with cognitive impairment AND past or present indication of BPSD, acutely admitted to the medicine or telemetry service, are cohorted on a 10-bed medical unit. II. PES staff. III. Staff Support: The PI will hold monthly 20 minute group sessions to reinforce training and discuss challenging patient behaviors; meant to improve the attitude and empathy of hospital caregivers towards patients. IV. Staff Training
  Interventions: Behavioral: PES-4-BPSD Model
- The attention control condition (Active Comparator): The control group consists of NAs that work on a 40-bed medicine unit, staffed with 39 nurses (1:6 ratio) and 26 NA (1:8 ratio), that primarily cohorts older patients with geriatric syndromes. All components of the intervention arm are the same with the exception of the PES staff. The control arm (NAs) will receive the same training as the intervention arm.
  Interventions: Behavioral: The attention control condition

INTERVENTIONS:
Behavioral: PES-4-BPSD Model — Staff Training: Dementia Care Education and Training. The PI, with the support of the research team, will spend 12 weeks training the PES/NA staff. Based on the "Try This: Best Practices in Nursing Care for Persons with Dementia," the PES staff will receive weekly 20 minute sessions. This study aims to capture the impact of dementia care training on the experience of PES (intervention unit) and NA (control unit) staff to care for patients with dementia. Measures will be completed at baseline, prior to dementia training (T1: baseline), immediately after completion of the training program (T2: 3 months post-baseline) and following the completion of the 1-year intervention period (T3: 12 months post-training).
  Arms: The PES-4-BPSD Model
Behavioral: The attention control condition — Staff Training: Dementia Care Education and Training. The PI, with the support of the research team, will spend 12 weeks to train the PES/NA staff. Based on the "Try This: Best Practices in Nursing Care for Persons with Dementia," the PES staff will receive weekly 20 minute sessions. This study aims to capture the impact of dementia care training on the experience of PES (intervention unit) and NA (control unit) staff to care for patients with dementia. Measures will be completed at baseline, prior to dementia training (T1: baseline), immediately after completion of the training program (T2: 3 months post-baseline) and following the completion of the 1-year intervention period (T3: 12 months post-training).
  Arms: The attention control condition

SUMMARY:
Persons with Alzheimer's Disease and Related Dementias (ADRD) account for 3.2 million hospital admissions per year and have over three times more hospitalizations than those without cognitive impairment, yet hospital caregivers (HCGs) are ill-prepared to manage patients with ADRD with less than 5% reporting mandatory dementia care training. Three-quarters of hospitalized persons with ADRD display Behavioral and Psychological Symptoms of Dementia (BPSD) associated with functional and cognitive decline, increased resource consumption, institutionalization, premature death, and caregiver burden. The overall objective is to test the preliminary efficacy of an innovative model of care, PES-4-BPSD, for reducing BPSD by empowering Patient Engagement Specialists (PES) to deliver dementia care for acutely-ill patients with ADRD. Traditionally, mental health assistants with training in crisis-prevention techniques provide care to psychiatric patients. On the intervention unit, these mental health assistants, as PES, purposefully engage patients with BPSD. In the pilot study, investigators found patients with cognitive impairment admitted to the PES unit were significantly less likely to require constant observation, chemical and physical restraints, suggesting improved management of BPSD. The central hypothesis is that PES-4-BPSD will improve the ability of PES to create an "enabling" milieu that addresses factors leading to BPSD and improves the experience of hospital caregivers. Guided by a social-ecological framework, PES-4-BPSD incorporates dementia education and training, environmental modifications-cohorting, increased staffing-PES, and staff support. The investigators' multidisciplinary research team is well-positioned to accomplish the following: Aim 1) Determine the preliminary efficacy of PES-4-BPSD for reducing BPSD during hospitalization (please refer to NCT# 04481568 for more details on this aim), and Aim 2) Evaluate whether dementia care training improves the perceived ability of PES staff (intervention) and nurse assistant staff (control) to care for hospitalized persons with ADRD. For Aim 1, investigators will conduct a non-randomized preliminary efficacy trial of the PES-4-BPSD intervention enrolling N=158 patients (79 control, 79 intervention). The primary outcome will be presence of BPSD during hospitalization using the Neuropsychiatric Inventory-Questionnaire (NPI-Q). In Aim 2, investigators will use survey methodology in a repeated measures design to evaluate within and between-group differences in attitudes, experience, and satisfaction toward managing patients with ADRD. Measures will be completed at baseline (T1), immediately following training (T2), and at the end of the intervention period (T3). This proposal will be the first to study an innovative model of care utilizing PES as specialized hospital caregivers for reducing BPSD in the hospital setting. The investigators' findings will lay the essential groundwork for a multi-site trial of PES-4-BPSD and inform the development of a program that can be easily implemented in other hospitals.

DETAILED DESCRIPTION:
We will evaluate whether dementia care training improves the perceived ability of PES staff (intervention) and nurse assistant staff (control) to care for hospitalized persons with ADRD. We will use survey methodology in a repeated measures design to evaluate within and between-group differences in attitudes, experience, and satisfaction toward managing patients with ADRD. Measures will be completed at baseline (T1), immediately following training (T2), and at end of the intervention period (T3). This study will utilize a repeated measures design to capture the impact of dementia care training on the experience of PES (intervention unit) and NA (control unit) staff to care for patients with dementia. Measures will be completed at baseline, prior to dementia training (T1: baseline), immediately after completion of the training program (T2: 3 months post-baseline) and following the completion of the 1-year intervention period (T3: 12 months post-training).

A 3 month dementia training program will be implemented on both the intervention and control units. On the intervention unit, training will target the PES and on the control to the nurse assistants. The 3 month dementia training program is based on the John A. Hartford Institute for Geriatric Nursing and the National Alzheimer Association publications Try This: Best Practices in Nursing Care for Persons with Dementia, "ACT" on Alzheimers guide to dementia friendly hospitals, and the Person-Centred Care Training Programme for Acute Hospitals (PCTAH), the research team will provide PES staff with weekly 20 minute sessions. The sessions will consists of the following topics: types and impact of dementia, providing person-centered care, identification of and meeting peoples emotional and physical needs, effective communication, connecting to the family caregiver (FCG), the impact of the physical environment, and redefining and supporting behaviors staff may describe as challenging. In order to ensure all staff get the training, sessions will be repeated 3 times per week during change of shift.

ELIGIBILITY:
Inclusion criteria:

* All PES staff on the intervention unit and nursing assistant staff on the control unit will be approached by research coordinator who has no authoritative responsibilities, emphasizing voluntary participation

Exclusion criteria:

* Staff who decline to participate in the study
* Staff that are not permanently based on either the intervention or control units

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liron Sinvani, MD, Principal Investigator — Northwell Health
Locations (2):
- United States (2):
  - Long Island Jewish Medical Center, Glen Oaks, New York
  - North Shore University Hospital, Manhasset, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sampson EL, White N, Leurent B, Scott S, Lord K, Round J, Jones L. Behavioural and psychiatric symptoms in people with dementia admitted to the acute hospital: prospective cohort study. Br J Psychiatry. 2014 Sep;205(3):189-96. doi: 10.1192/bjp.bp.113.130948. Epub 2014 Jul 24. PMID 25061120
- [Background] Hessler JB, Schaufele M, Hendlmeier I, Junge MN, Leonhardt S, Weber J, Bickel H. Behavioural and psychological symptoms in general hospital patients with dementia, distress for nursing staff and complications in care: results of the General Hospital Study. Epidemiol Psychiatr Sci. 2018 Jun;27(3):278-287. doi: 10.1017/S2045796016001098. Epub 2017 Jan 9. PMID 28065176
- [Background] Astrom S, Nilsson M, Norberg A, Sandman PO, Winblad B. Staff burnout in dementia care--relations to empathy and attitudes. Int J Nurs Stud. 1991;28(1):65-75. doi: 10.1016/0020-7489(91)90051-4. PMID 1856035
- [Background] Dewing J, Dijk S. What is the current state of care for older people with dementia in general hospitals? A literature review. Dementia (London). 2016 Jan;15(1):106-24. doi: 10.1177/1471301213520172. Epub 2014 Jan 23. PMID 24459188
- [Background] Lintern TC. Quality in dementia care: evaluating staff attitudes and behaviour. [PhD Thesis]. Prifysgol Bangor University; 2001.
- [Background] Scerri A, Innes A, Scerri C. Dementia training programmes for staff working in general hospital settings - a systematic review of the literature. Aging Ment Health. 2017 Aug;21(8):783-796. doi: 10.1080/13607863.2016.1231170. Epub 2016 Sep 23. PMID 27662075
- [Result] Sinvani L, Warner-Cohen J, Strunk A, Halbert T, Harisingani R, Mulvany C, Qiu M, Kozikowski A, Patel V, Liberman T, Carney M, Pekmezaris R, Wolf-Klein G, Karlin-Zysman C. A Multicomponent Model to Improve Hospital Care of Older Adults with Cognitive Impairment: A Propensity Score-Matched Analysis. J Am Geriatr Soc. 2018 Sep;66(9):1700-1707. doi: 10.1111/jgs.15452. Epub 2018 Aug 11. PMID 30098015
- See also: Please refer to NCT# 04481568 for more details on Aim 1: Family Caregivers — https://clinicaltrials.gov/ct2/show/NCT04481568

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | The PES-4-BPSD Model | The Attention Control Condition
Started (Enrolled) | 22 | 32
T1 - Baseline | 16 | 24
T2 - Post-Training | 16 | 21
T3 - End of Intervention | 11 | 18
Completed | 11 | 18
Not Completed | 11 | 14
Not completed — COVID-19 Related Lost of Followup | 11 | 13
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | The PES-4-BPSD Model | The Attention Control Condition | Total
Number analyzed (Participants) | 22 | 32 | 54
Age, Customized [Count of Participants; unit: Participants]
  18-24 years | 1 | 5 | 6
  25-34 years | 6 | 12 | 18
  35-44 years | 10 | 3 | 13
  45-54 years | 2 | 6 | 8
  55-64 years | 3 | 4 | 7
  65-74 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 26 | 42
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 20 | 27 | 47
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 20 | 35
  White | 2 | 5 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 5 | 7
Years Working in Acute Care [Count of Participants; unit: Participants]
  0-5 years | 5 | 15 | 20
  6-10 years | 11 | 6 | 17
  11-15 years | 2 | 3 | 5
  16-20 years | 2 | 3 | 5
  > 20 years | 2 | 5 | 7
Shift [Count of Participants; unit: Participants]
  Day | 7 | 14 | 21
  Evening | 10 | 9 | 19
  Night | 5 | 9 | 14
Previous Dementia Training/Education [Count of Participants; unit: Participants]
  None | 8 | 26 | 34
  1-2 Hours | 4 | 3 | 7
  Half Day | 3 | 0 | 3
  Full Day | 2 | 0 | 2
  Other | 5 | 2 | 7
  Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Approaches to Dementia Questionnaire (ADQ) Total Score From Baseline to 3 Months
Description: The Approaches to Dementia Questionnaire (ADQ) is a 19-item scale designed to evaluate staff attitudes to people with dementia and providing dementia care. A five-point Likert Scale (1-5) is used for each item. The ADQ total score ranges from 19-95 with higher scores indicating a more positive attitude. The ADQ will be completed by Patient Engagement Specialists and Nurse Assistants at baseline (enrollment) and 3 months from enrollment. The average ADQ score at baseline and at 3 months was calculated separately for each group and change was assessed by subtracting each group's average score at their respective timepoints. Missing values for each item were imputed using the group mode for that item. 95% confidence intervals were calculated based on the t-distribution assuming independence of observations across time periods. Paired analysis was not feasible given anonymous data.
Time Frame: Baseline and 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | The PES-4-BPSD Model | The Attention Control Condition
Number analyzed (Participants) | 22 | 32
units on a scale | -1.8 [-6.3 to 2.6] | -2.3 [-6.3 to 1.7]

2. Primary Outcome: Change in Staff Experiences of Working With Demented Residents Scale Total Score From Baseline to 3 Months
Description: The Staff Experience of Working with Demented Residents Scale (SEWDR) is a 21-item scale measuring staff satisfaction in their work environment and working with people with dementia. A five-point Likert scale (0-4) is used for each item. The SEWDR total score ranges from 0-84; higher scores indicate greater satisfaction. Patient Engagement Specialists and Nurse Assistants will complete the SEWDR at baseline (enrollment) and 3 months from enrollment. The average score at baseline and at 3 months will be calculated separately for each group; change will be assessed by subtracting each group's average score at their respective timepoints. Missing values for each item were imputed using the group mode for that item. 95% confidence intervals were calculated based on the t-distribution assuming independence of observations across time periods. Paired analysis was not feasible given anonymous data.
Time Frame: Baseline and 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | The PES-4-BPSD Model | The Attention Control Condition
Number analyzed (Participants) | 22 | 32
units on a scale | 2.9 [-3.6 to 9.3] | 4.0 [-0.9 to 9.0]

3. Primary Outcome: Change in Approaches to Dementia Questionnaire (ADQ) Total Score From Baseline to 15 Months
Description: The Approaches to Dementia Questionnaire (ADQ) is a 19-item scale designed to evaluate staff attitudes to people with dementia and providing dementia care. A five-point Likert Scale (1-5) is used for each item. The ADQ total score ranges from 19-95 with higher scores indicating a more positive attitude. The ADQ will be completed by Patient Engagement Specialists and Nurse Assistants at baseline (enrollment) and 15 months from enrollment. The average ADQ score at baseline and at 15 months was calculated separately for each group and change was assessed by subtracting each group's average score at their respective timepoints. Missing values for each item were imputed using the group mode for that item. 95% confidence intervals were calculated based on the t-distribution assuming independence of observations across time periods. Paired analysis was not feasible given anonymous data.
Time Frame: Baseline and 15 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | The PES-4-BPSD Model | The Attention Control Condition
Number analyzed (Participants) | 22 | 32
units on a scale | -0.9 [-5.8 to 4.1] | -4.5 [-8.7 to -0.3]

4. Primary Outcome: Change in Staff Experiences of Working With Demented Residents Scale Total Score From Baseline to 15 Months
Description: The Staff Experience of Working with Demented Residents Scale (SEWDR) is a 21-item scale measuring staff satisfaction in their work environment and working with people with dementia. A five-point Likert scale (0-4) is used for each item. The SEWDR total score ranges from 0-84; higher scores indicate greater satisfaction. Patient Engagement Specialists and Nurse Assistants will complete the SEWDR at baseline (enrollment) and 15 months from enrollment. The average score at baseline and at 15 months will be calculated separately for each group; change will be assessed by subtracting each group's average score at their respective timepoints. Missing values for each item were imputed using the group mode for that item. 95% confidence intervals were calculated based on the t-distribution assuming independence of observations across time periods. Paired analysis was not feasible given anonymous data.
Time Frame: Baseline and 15 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | The PES-4-BPSD Model | The Attention Control Condition
Number analyzed (Participants) | 22 | 32
units on a scale | 4.8 [-3.7 to 13.2] | 0.9 [-5.0 to 6.7]

5. Secondary Outcome: Approaches to Dementia Questionnaire Total Score at Baseline
Description: The Approaches to Dementia Questionnaire (ADQ) is a 19-item scale designed to evaluate staff attitudes to people with dementia and providing dementia care. A five-point Likert Scale (1 to 5) is used for each survey item. The total score for the ADQ ranges from 19 to 95, with higher scores indicating a more positive attitude. The ADQ will be completed by Patient Engagement Specialist (PES) staff and Nurse Assistant (NA) staff at enrollment (baseline), and mean score will be compared between these groups.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The PES-4-BPSD Model | The Attention Control Condition
Number analyzed (Participants) | 22 | 32
score on a scale | 70.3 (6.4) | 69.2 (6.5)

6. Secondary Outcome: Staff Experiences of Working With Demented Residents Scale Total Score at Baseline
Description: The Staff Experience of Working with Demented Residents Scale (SEWDR) is a 21-item scale measuring staff satisfaction in their experiences working with people with dementia as well as their work environment. A five-point Likert scale (0 to 4) is used for each survey item. The total score for the SEWDR ranges from 0 to 84, with higher scores indicating greater satisfaction. The SEWDR will be completed by Patient Engagement Specialist (PES) staff and Nurse Assistant (NA) staff at enrollment (baseline), and mean score will be compared between these groups.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The PES-4-BPSD Model | The Attention Control Condition
Number analyzed (Participants) | 22 | 32
score on a scale | 52.2 (10.1) | 50.8 (10.2)

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | The PES-4-BPSD Model | The Attention Control Condition
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/32
Other Adverse Events (participants affected / at risk) | 0/22 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT04179721/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT04179721/ICF_001.pdf